CLINICAL TRIAL: NCT04328077
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2a Clinical Trial to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Orally Administered TERN-101 Tablets in Adult Patients With Presumed Non-Cirrhotic Non-Alcoholic Steatohepatitis (NASH)
Brief Title: LIFT Study: A Safety, Tolerability, Efficacy, and Pharmacokinetics Study of TERN-101 in Subjects With Non-Cirrhotic Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Terns, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TERN101-2001
Record Dates: First submitted 2020-03-13; First posted 2020-03-31 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Farnesoid X receptor; NASH; Nonalcoholic Steatohepatitis; NAFLD; Nonalcoholic Fatty Liver Disease; FXR
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TERN-101 dose level 1 (Experimental): Orally administered.
  Interventions: Drug: TERN-101
- TERN-101 dose level 2 (Experimental): Orally administered.
  Interventions: Drug: TERN-101
- TERN-101 dose level 3 (Experimental): Orally administered.
  Interventions: Drug: TERN-101
- Placebo (Placebo Comparator): Orally administered.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TERN-101 — Investigational drug
  Arms: TERN-101 dose level 1; TERN-101 dose level 2; TERN-101 dose level 3
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, efficacy, and pharmacokinetics (PK) of TERN-101 in non-cirrhotic NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Overweight or obese with a body mass index (BMI) ≥ 25 kg/m2
* Presumed NASH based on clinical characteristics or prior liver biopsy
* ALT ≥ 43 IU/L for men and ≥ 28 IU/L for women
* MRI PDFF liver fat content ≥ 10 %
* Written informed consent

Exclusion Criteria:

* History or clinical evidence of chronic liver diseases other than NAFLD
* History or clinical evidence of cirrhosis, hepatic decompensation or other severe liver impairment
* History of liver transplant, or current placement on a liver transplant list
* Total bilirubin > 1.2 mg/dL
* Albumin < 3.5 g/dL
* INR > 1.1
* AST or ALT > 5 x ULN
* ALP > 156 IU/L
* Platelet count < 150,000 /mm3
* eGFR < 60 mL/min/1.73m2
* Weight loss > 5% within past 3 months prior to Screening
* Uncontrolled diabetes
* Uncontrolled hyperlipidemia
* Active COVID-19 infection
* Other protocol-defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: clinicaltrials@ternspharma.com, Study Director — Terns, Inc.
Locations (31):
- United States (31):
  - Terns Clinical Study Site 1017, Chandler, Arizona
  - Terns Clinical Study Site 1018, Tucson, Arizona
  - Terns Clinical Study Site 1024, Tucson, Arizona
  - Terns Clinical Study Site 1004, Coronado, California
  - Terns Clinical Study Site 1035, Fresno, California
  - Terns Clinical Study Site 1013, La Jolla, California
  - Terns Clinical Study Site 1016, Los Angeles, California
  - Terns Clinical Study Site 1008, Montclair, California
  - Terns Clinical Study Site 1001, Panorama City, California
  - Terns Clinical Study Site 1012, Gainesville, Florida
  - Terns Clinical Study Site 1007, Hialeah, Florida
  - Terns Clinical Study Site 1028, Hialeah, Florida
  - Terns Clinical Study Site 1009, Miami, Florida
  - Terns Clinical Study Site 1033, Orlando, Florida
  - Terns Clinical Study Site 1032, Indianapolis, Indiana
  - Terns Clinical Study Site 1010, Bastrop, Louisiana
  - Terns Clinical Study Site 1037, New Orleans, Louisiana
  - Terns Clinical Study Site 1023, Shreveport, Louisiana
  - Terns Clinical Study Site 1002, Baltimore, Maryland
  - Terns Clinical Study Site 1011, Boston, Massachusetts
  - Terns Clinical Study Site 1038, Florham Park, New Jersey
  - Terns Clinical Study Site 1027, Durham, North Carolina
  - Terns Clinical Study Site 1014, Hermitage, Tennessee
  - Terns Clinical Study Site 1005, Arlington, Texas
  - Terns Clinical Study Site 1025, Georgetown, Texas
  - Terns Clinical Study Site 1021, Houston, Texas
  - Terns Clinical Study Site 1029, Houston, Texas
  - Terns Clinical Study Site 1006, San Antonio, Texas
  - Terns Clinical Study Site 1003, San Antonio, Texas
  - Terns Clinical Study Site 1019, San Antonio, Texas
  - Terns Clinical Study Site 1022, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Comparator: Placebo: Orally administered
- TERN-101 5mg: Experimental: TERN-101 dose level 1: Orally administered
- TERN-101 10mg: Experimental: TERN-101 dose level 2: Orally administered
- TERN-101 15mg: Experimental: TERN-101 dose level 3: Orally administered
Period: Overall Study
Arm/Group | Placebo | TERN-101 5mg | TERN-101 10mg | TERN-101 15mg
Started | 26 | 25 | 26 | 24
Completed | 26 | 23 | 25 | 21
Not Completed | 0 | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TERN-101 5mg | TERN-101 10mg | TERN-101 15mg | Total
Number analyzed (Participants) | 26 | 25 | 26 | 23 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 23 | 21 | 94
  >=65 years | 0 | 1 | 3 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (11.00) | 48.0 (12.32) | 52.5 (13.64) | 51.6 (9.49) | 50.6 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 17 | 17 | 65
  Male | 10 | 10 | 9 | 6 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 23 | 21 | 21 | 86
  Black or African American | 2 | 1 | 2 | 0 | 5
  Asian | 1 | 1 | 1 | 0 | 3
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 2 | 0 | 2 | 2 | 6
  Unknown | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 17 | 16 | 17 | 70
  Not Hispanic or Latino | 6 | 8 | 9 | 4 | 27
  Not Reported | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 26 | 23 | 100
ALT [Mean (Standard Deviation); unit: U/L] — Baseline ALT (U/L) was defined as the average of all assessments prior to dosing.
  U/L | 55.51 (23.639) | 56.25 (16.266) | 60.84 (29.075) | 55.79 (26.447) | 57.15 (24.064)
Diabetes Mellitus Status [Count of Participants; unit: Participants] — Diabetes Mellitus status was defined as having reported any medical history MedDRA preferred term including "Diabetes mellitus" or "Diabetic neuropathy" or "Diabetic retinopathy".
  Participants
    Absent | 15 | 14 | 10 | 15 | 54
    Present | 11 | 11 | 16 | 8 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events for TERN-101 Versus Placebo
Time Frame: 16 weeks
Population: Safety Population: All patients who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- TERN-101 5 mg: Experimental: TERN-101 dose level 1: Orally administered
- TERN-101 10 mg: Experimental: TERN-101 dose level 2: Orally administered
- TERN-101 15 mg: Experimental: TERN-101 dose level 3: Orally administered
Arm/Group | Placebo | TERN-101 5 mg | TERN-101 10 mg | TERN-101 15 mg
Number analyzed (Participants) | 26 | 25 | 26 | 23
Participants | 10 | 13 | 14 | 15

2. Secondary Outcome: Percent Change From Baseline in ALT Outcome Measure
Time Frame: 12 weeks
Population: Efficacy Population: All randomized patients who received at least 1 dose of study drug
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Placebo | TERN-101 5 mg | TERN-101 10 mg | TERN-101 15 mg
Number analyzed (Participants) | 25 | 24 | 25 | 21
percentage of change from baseline | -5.33 (6.606) | -2.63 (6.743) | -17.99 (6.646) | -13.22 (7.246)
Statistical Analysis 1: Comparison: Placebo vs TERN-101 5 mg; Test type: Superiority; p = 0.7755, ANCOVA; Mean Difference (Final Values) = 2.70, 95% CI 2-sided [-16.1 to 21.5], Standard Error of Mean 9.440
Statistical Analysis 2: Comparison: Placebo vs TERN-101 10 mg; Test type: Superiority; p = 0.1798, ANCOVA; Mean Difference (Final Values) = -12.66, 95% CI 2-sided [-31.3 to 5.9], Standard Error of Mean 9.369
Statistical Analysis 3: Comparison: Placebo vs TERN-101 15 mg; Test type: Superiority; p = 0.4229, ANCOVA; Mean Difference (Final Values) = -7.90, 95% CI 2-sided [-27.4 to 11.6], Standard Error of Mean 9.807

3. Secondary Outcome: Plasma Concentration of TERN-101 - AUC 0-24
Description: Area under the curve
Time Frame: 12 weeks (0-24 hours post dose)
Population: All randomized patients in the PK/PD substudy who received at least 1 dose of TERN-101. The minimum requirement for the calculation of AUC required: A minimum of 3 measurable concentration-time-points during the log-linear portion of the terminal elimination phase (after tmax), excluding Cmax; r²adj ≥ 0.80 for the regression of the log-concentration time data during the terminal elimination phase; Negative slope for log regression fit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TERN-101 5mg | TERN-101 10mg | TERN-101 15mg
Number analyzed (Participants) | 4 | 4 | 5
h*ng/mL | 1380 (96.7) | 1470 (29.7) | 2510 (13.3)

4. Secondary Outcome: Plasma Concentration of TERN-101 - Cmax
Description: Maximum observed concentration
Time Frame: 12 Weeks (0-72 hours post dose)
Population: All randomized patients in the PK/PD substudy who received at least 1 dose of TERN-101.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TERN-101 5 mg | TERN-101 10 mg | TERN-101 15 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 116 (45.0) | 155 (158.8) | 389 (19.0)

5. Secondary Outcome: Plasma Concentration of TERN-101 - Tmax
Description: Time to reach maximum measured plasma concentration
Time Frame: 12 Weeks (0-72 hours post dose)
Population: All randomized patients in the PK/PD substudy who received at least 1 dose of TERN-101.
Measure: Median (Full Range); unit: hour
Arm/Group | TERN-101 5 mg | TERN-101 10 mg | TERN-101 15 mg
Number analyzed (Participants) | 6 | 6 | 6
hour | 1 [0 to 6] | 1 [0 to 3] | 0.5 [0.5 to 1]

6. Secondary Outcome: Plasma Concentration of TERN-101 - t1/2
Description: Determination of half-life
Time Frame: 12 Weeks (0-72 hours post dose)
Population: All randomized patients in the PK/PD substudy who received at least 1 dose of TERN-101. The minimum requirement for the calculation of t1/2 required: A minimum of 3 measurable concentration-time-points during the log-linear portion of the terminal elimination phase (after Tmax), excluding Cmax; r²adj ≥ 0.80 for the regression of the log-concentration time data during the terminal elimination phase; and negative slope for log regression fit.
Measure: Median (Full Range); unit: hour
Arm/Group | TERN-101 5 mg | TERN-101 10 mg | TERN-101 15 mg
Number analyzed (Participants) | 4 | 4 | 5
hour | 14.6 [8.7 to 67.8] | 6.75 [4 to 7.9] | 6 [5.8 to 11.3]

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | Placebo | TERN-101 5mg | TERN-101 10mg | TERN-101 15mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/25 | 0/26 | 1/23
Other Adverse Events (participants affected / at risk) | 10/26 | 13/25 | 14/26 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | TERN-101 5mg (N=25) | TERN-101 10mg (N=26) | TERN-101 15mg (N=23)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | TERN-101 5mg (N=25) | TERN-101 10mg (N=26) | TERN-101 15mg (N=23)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Magnetic resonance imaging abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04328077/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT04328077/SAP_001.pdf